CLINICAL TRIAL: NCT03526016
Title: Effect of Transsphenoidal Surgery on Sleep Apnea in Patients With Acromegaly
Brief Title: Sleep Apnea in Acromegaly After Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Associate professor, Seoul National University Hospital
Other Study IDs: 1802032919
Record Dates: First submitted 2018-05-02; First posted 2018-05-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Sleep Apnea
Keywords: Sleep Apnea; Acromegaly; Transsphenoidal surgery; Respiratory polygraphy
MeSH Terms: conditions — Sleep Apnea Syndromes; Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep apnea is common in acromegaly and both diseases are independently associated with hypertension and insulin resistance contributing to increased morbidity and mortality. Respiratory polygraphy is a simpler alternative to in-laboratory polysomnography for the management of more symptomatic patients with obstructive sleep apnea.

The aim of this study is to evaluate the prevalence of sleep apnea by respiratory polygraphy, and to analyze the effect of transsphenoidal surgery on sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed acromegaly

Exclusion Criteria:

* patients who can not undergo transsphenoidal surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Respiratory disturbance index | Baseline and 3 months after transsphenoidal surgery
  Changes in respiratory events during sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho J, Kim JH, Kim YH, Lee J. Obstructive Sleep Apnea Screening and Effects of Surgery in Acromegaly: A Prospective Study. Endocrinol Metab (Seoul). 2024 Aug;39(4):641-652. doi: 10.3803/EnM.2024.1933. Epub 2024 Jun 26. PMID 38918903